CLINICAL TRIAL: NCT04984850
Title: Feasibility, Acceptability, and Potential Effects of a Comprehensive Oral Chemotherapy Intervention on Medication Adherence Self-efficacy, Medication Adherence, and Symptom Distress: A Pilot Randomized Control Trial
Brief Title: Oncology - Bolstering Oral Agent Reporting Related to Distress
Acronym: ON-BOARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Rossy Cancer Network (Unknown)
Responsible Party: Principal Investigator, Carmen G. Loiselle, N., Ph.D., Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-2861
Record Dates: First submitted 2021-06-09; First posted 2021-08-02 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Oral Chemotherapy
Keywords: Oral chemotherapy; medication adherence; self-efficacy; pilot randomized control trial
MeSH Terms: conditions — Medication Adherence | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Following baseline, participants randomized immediately to receive either the intervention plus usual care (experimental group, n = 26) or usual care only (control group, n = 26).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention plus usual care (Experimental)
  Interventions: Other: Oral chemotherapy information and support
- Usual care only (No Intervention)

INTERVENTIONS:
Other: Oral chemotherapy information and support — Multimodal intervention : (1) handouts and videos presenting information and supportive resources for common oral chemotherapy related issues, (2) phone call(s) from a nurse in oncology, and (3) e-reminders to take medication. The intervention will be available to experimental group participants on mobile platform.
  Arms: Intervention plus usual care

SUMMARY:
Individuals on oral chemotherapy (OC) often face many challenges requiring adequate informational support, monitoring, and management. This pilot randomized control trial (RCT) aims to assess the feasibility, acceptability, and preliminary effects of a comprehensive OC intervention on medication adherence self-efficacy, medication adherence, and symptom distress.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of cancer, any stage
* Being followed by a care team at the affiliated hospital centre
* About to start or within the first cycle of oral anticancer treatment (traditional cytotoxic, targeted therapy, hormonal therapy as active ongoing treatment for cancer with the aim of killing cancer cells/shrinking tumor size)
* Has a computer/tablet/smartphone device with internet
* The ability to communicate, read, and write in English or French

Exclusion Criteria:

* Receiving IV chemotherapy, immunotherapy, and/or oral hormonal therapy as long-term maintenance treatment for prevention of cancer's return/growth of cancer cells after initial treatment
* Significant physical or cognitive limitations that would prevent ability to participate in study as reported by patient, primary healthcare provider, or research staff
* At imminent "end-of-life"
* Participating in an ongoing clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability | Five months
  Study feasibility assessed by the recruitment rate (percentage, dividing the total number of participants recruited throughout the study by the number of months recruitment occurred), retention rate (percentage, comparing the number of participants who complete baseline e-questionnaires to the number of participants who complete study exit e-questionnaires), response rate to study e-questionnaires (percentage, the number of completed follow-up e-questionnaire assessments for participants who complete the study), and uptake of intervention (percentage, calculated by comparing by number of participants who actually access the intervention to the total number who are given access).
  Intervention acceptability assessed by intervention burden, intervention coherence, and perceived effectiveness using the Tariman et al. (2011) Acceptability e-scale for web-based patient-reported outcomes in cancer care. Mean scores range from 1 to 5, higher score indicating higher acceptability.

SECONDARY OUTCOMES:
Potential effects of intervention via medication adherence self-efficacy, medication adherence and symptom distress | Five months
  Medication adherence self-efficacy by the Medication Adherence Self-Efficacy Scale (MASES) (Ogedegbe et al., 2003). Total scores range from 20 to 60, higher scores indicating higher medication adherence self-efficacy.
  Medication adherence via Proportion of Days Covered (PDC), percentage representing the sum of the days' supply of a given drug divided by the number of days in the time period. Higher percentage indicating higher medication adherence.
  Medication adherence self-report via the Medication Adherence Report Scale (MARS-5, Professor Rob Horne; Chan et al., 2020). Total scores range from 5 to 25, higher score indicating higher self-reported adherence.
  Physical and psychosocial symptom distress measured via Edmonton Symptom Assessment Scale Revised (ESAS-r) for anxiety, depression, drowsiness, fatigue, fear of cancer recurrence, lack of appetite, nausea, shortness of breath, sleep, wellbeing, and work. Each is rated from 0 to 10, 0 being none and 10 being the worst possible.

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS du Centre-Ouest-de-l'Île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed S, Maheu C, Gotlieb W, Batist G, Loiselle CG. Feasibility, Acceptability, and Potential Effects of a Digital Oral Anticancer Agent Intervention: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 26;14:e55475. doi: 10.2196/55475. PMID 40138678